CLINICAL TRIAL: NCT02657928
Title: A Phase 2 Trial of Ribociclib (LEE011) and Letrozole in ER Positive Relapsed Ovarian Cancer, Fallopian Tube Cancer, Primary Peritoneal Carcinomas, and Endometrial Cancers.
Brief Title: Ribociclib and Letrozole in Treating Patients With Relapsed ER Positive Ovarian, Fallopian Tube, Primary Peritoneal, or Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1561; NCI-2015-02181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1561 (Other: Mayo Clinic in Florida); P30CA015083 (NIH)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Estrogen Receptor Positive; Postmenopausal; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Letrozole; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ribociclib and letrozole) (Experimental): Patients receive ribociclib PO daily and letrozole PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Letrozole; Drug: Ribociclib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Ribociclib — Given PO
  Other Names: LEE-011; LEE011

SUMMARY:
This phase II trial studies how well ribociclib and letrozole work in treating patients with estrogen receptor (ER) positive ovarian, fallopian tube, primary peritoneal, or endometrial cancer that has returned (come back) after a period of improvement. Ribociclib may stop the growth of tumor cells by blocking some enzymes needed for cell growth. Cancer cells that are estrogen receptor positive may need estrogen to grow. Letrozole lowers the amount of estrogen made by the body and this may stop the growth of tumor cells that need estrogen to grow. Giving ribociclib together with letrozole may be an effective treatment in patients with ovarian, fallopian tube, primary peritoneal, or endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate if the combination of letrozole and ribociclib (LEE011) leads to a higher percentage of patients who are progression free at 12 weeks (PFS 12) as compared with that observed in prior studies with single agent letrozole.

SECONDARY OBJECTIVES:

I. Demonstrate if the combination of letrozole and ribociclib (LEE011) leads to a higher cancer antigen 125 (CA-125) response rate in patients with relapsed ER positive ovarian cancers and endometrial cancers as compared to that observed in previously reported single agent letrozole studies.

II. Median progression-free survival (PFS), overall survival (OS), the confirmed response rate, and adverse events.

TERTIARY OBJECTIVES:

I. Identify molecular biomarkers associated with a response to treatment with letrozole and ribociclib (LEE011) (in patients with relapsed ovarian carcinomas and endometrial cancers).

II. Develop patient derived xenograft (PDX) avatars on tumors from participants for possible future translational study evaluating a potential correlation between responses in the PDX model to patients' responses.

OUTLINE:

Patients receive ribociclib orally (PO) daily and letrozole PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Post-menopausal
* Histologically confirmed recurrent ovarian, fallopian tube or primary peritoneal carcinoma or endometrial cancer in post-menopausal women; NOTE: pure clear cell and pure mucinous carcinomas are ineligible; platinum sensitive, platinum resistant and platinum refractory disease are eligible; no limitations in the number of prior regimens
* Patient has disease amenable to biopsy and is agreeable to undergo a biopsy; NOTE: under unusual circumstances, submission of ascites material may be acceptable if a biopsy is not possible; this exception will require approval by one of the study principal investigators
* Willing to provide tissue samples for ER and retinoblastoma (RB) staining
* Measurable disease by Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Tumors must stain positive for estrogen receptor (>= 10%) by immunohistochemistry (IHC)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1 x upper limit of normal (ULN); or total bilirubin =< 3.0 x ULN with direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome
* Aspartate transaminase (aspartate aminotransferase [AST]) =< 2.5 x ULN (=< 5 x ULN in patients with liver metastasis)
* International normalized ratio (INR) =< 2
* Creatinine =< 1.5 mg/dL
* Potassium =< ULN (or corrected to =< ULN with supplements prior to registration)
* Total calcium (corrected for serum calcium) =< ULN (or corrected to =< ULN with supplements prior to registration)
* Magnesium =< ULN (or corrected to =< ULN with supplements prior to registration)
* Sodium =< ULN (or corrected to =< ULN with supplements prior to registration)
* Phosphorus =< ULN (or corrected to =< ULN with supplements prior to registration)
* Ability to swallow study medication
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide tissue samples for correlative research purposes

Exclusion Criteria:

* Patients who have central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * >= 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.)
* Clinically significant, uncontrolled heart disease or cardiac repolarization abnormalities and/or recent events including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
  * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g. bifascicular block, Mobitz type II and third-degree AV block) long QT syndrome or family history of long QT syndrome
  * Idiopathic sudden death or congenital long QT syndrome
  * Risk factors for torsades de pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause torsades de pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
  * Inability to determine the QT interval on screening (corrected QT interval [QTcF], using Fridericia's correction)
  * Systolic blood pressure (SBP) > 160 mmHg or < 90 mmHg at screening
  * Bradycardia (heart rate < 50 at rest), by electrocardiogram (ECG) or pulse, at screening
  * Tachycardia (heart rate > 110 at rest), by ECG or pulse at screening
* Inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF > 450 msec (using Fridericia's correction); NOTE: all as determined by screening ECG
* Patient is currently receiving any of the following medications and cannot be discontinued =< 7 days prior to starting study drug: known strong inducers or inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4/5 (CYP3A4/5) including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges or that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5 or herbal preparations/medications or dietary supplements
* Patient is currently receiving or has received systemic corticosteroids within =< 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment; NOTE: the following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patient has received radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom >= 30% of the bone marrow was irradiated
* Patient has had major surgery =< 14 days prior to registration or has not recovered from major side effects (tumor biopsy is not considered as major surgery)
* Known to be human immunodeficiency virus (HIV) positive (testing not mandatory)
* Patient has a known hypersensitivity to any of the excipients of ribociclib
* Patient is currently receiving warfarin or other Coumarin-derived anticoagulant for treatment, prophylaxis or otherwise; NOTE: therapy with apixaban, dabigatran, heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed
* Participation in a prior investigational study within 30 days prior to enrollment or =< 5 half-lives of the investigational product, whichever is longer
* Patient has not recovered from all toxicities related to prior anticancer therapies to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 grade < 3 (exception to this criterion: patients with any grade of alopecia or neuropathy are allowed to enter the study)
* Patient with a Child-Pugh score B or C
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or significant small bowel resection)
* Prior therapy with ribociclib or an aromatase inhibitor (letrozole, anastrozole or exemestane)
* Patient has received systemic chemotherapy =< 3 weeks prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Colon-Otero, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Colon-Otero G, Zanfagnin V, Hou X, Foster NR, Asmus EJ, Wahner Hendrickson A, Jatoi A, Block MS, Langstraat CL, Glaser GE, Dinh TA, Robertson MW, Camoriano JK, Butler KA, Copland JA, Weroha SJ. Phase II trial of ribociclib and letrozole in patients with relapsed oestrogen receptor-positive ovarian or endometrial cancers. ESMO Open. 2020 Oct;5(5):e000926. doi: 10.1136/esmoopen-2020-000926. PMID 33109627

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Ovarian: Patients with ovarian, primary peritoneal, fallopian tube ACA receive ribociclib 400 mg PO daily and letrozole 2.5 mg PO daily on days 1-28.
- Cohort B: Endometrial: Patients with endometrial cancer receive ribociclib 400 mg PO daily and letrozole 2.5 mg PO daily on days 1-28.
Period: Overall Study
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 82] | 64.5 [52 to 75] | 64 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 12 | 11 | 23
    1 | 7 | 6 | 13
    2 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Free of Progression at 12 Weeks (PFS12)
Description: The percentage of patients who are progression-free at 12 weeks (PFS12) is defined as patients who are alive and progression free at 12 weeks. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: At 12 weeks
Population: Per protocol analysis population: 19 evaluable patients per cohort
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
Number analyzed (Participants) | 19 | 19
percentage of patients | 52.6 | 57.9

2. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of registration to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: From registration to the first of either disease progression or death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
Number analyzed (Participants) | 20 | 20
months | 2.8 [2.6 to 9.1] | 5.4 [3.1 to 11.8]
Statistical Analysis 1: Comparison: Cohort A: Ovarian vs Cohort B: Endometrial; Test type: Superiority; p = 0.5004, Log Rank

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: From registration to death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
Number analyzed (Participants) | 20 | 20
months | 18.9 [6.7 to NA] — The 95% confidence interval upper limit was not evaluated (below the level of detection). | 15.7 [6.8 to NA] — The 95% confidence interval upper limit was not evaluated (below the level of detection).
Statistical Analysis 1: Comparison: Cohort A: Ovarian vs Cohort B: Endometrial; Test type: Superiority; p = 0.9127, Log Rank

4. Secondary Outcome: The Number of Patients With CA-125 Response
Description: The number of patients with CA-125 response, defined as a 50% or greater reduction in baseline CA-125.
Time Frame: Up to 2 years
Population: Patients with CA-125 response data available with abnormal values at baseline are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Overall (Cohort A + Cohort B): Patients with either ovarian, primary peritoneal, fallopian tube ACA or endometrial cancer receive ribociclib 400 mg PO daily and letrozole 2.5 mg PO daily on days 1-28.
Arm/Group | Overall (Cohort A + Cohort B)
Number analyzed (Participants) | 27
Participants | 4

5. Secondary Outcome: The Number of Patients With Confirmed Response (Complete Response or Partial Response)
Description: The number of patients with confirmed response (complete response or partial response) using Response Evaluation Criteria in Solid Tumors version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
Number analyzed (Participants) | 20 | 20
Participants | 3 | 3

6. Secondary Outcome: The Number of Treatment-related Grade 3 or Higher Adverse Events
Description: The number of treatment-related Grade 3 or higher adverse events using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to 30 days post-treatment
Measure: Number; unit: events
Arm/Group | Overall (Cohort A + Cohort B)
Number analyzed (Participants) | 40
events
  Grade 3 : Lymphopenia | 5
  Grade 3 : Leukopenia | 8
  Grade 3 : Neutropenia | 6
  Grade 3 : Febrile Neutropenia | 0
  Grade 3 : Fatigue | 2
  Grade 3 : Liver Enzymes | 3
  Grade 4 : Lymphopenia | 1
  Grade 4 : Leukopenia | 0
  Grade 4 : Neutropenia | 0
  Grade 4 : Febrile Neutropenia | 1
  Grade 4 : Fatigue | 0
  Grade 4 : Liver Enzymes | 0

7. Other Pre Specified Outcome: Creation of Patient Derived Xenograft Models for Future Translational Experiments
Description: Xenograft will be created on each patient. For patient derived xenograft experiments, response to therapy will be based on tumor volumes measured by ultrasound. Tumor growth curves will be plotted graphically and notated to indicate the outcome status of the originating patients. End of study tumor volumes will be correlated with outcome status of the originating patient as well.
Time Frame: 28 days following treatment initiation
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Molecular Biomarkers Associated With a Response to Treatment With Letrozole and Ribociclib
Description: Whether response rates to letrozole and ribociclib in patient derived xenograft avatars correlate to responses noted in the patients will be determined. Fisher's Exact test will be used to measure the associations.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days post-treatment
Arm/Group | Cohort A: Ovarian | Cohort B: Endometrial
All-Cause Mortality (participants affected / at risk) | 10/20 | 10/20
Serious Adverse Events (participants affected / at risk) | 6/20 | 10/20
Other Adverse Events (participants affected / at risk) | 18/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Ovarian (N=20) | Cohort B: Endometrial (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Ovarian (N=20) | Cohort B: Endometrial (N=20)
Anemia (Blood and lymphatic system disorders) | 7 (25) | 5 (23)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (6)
Constipation (Gastrointestinal disorders) | 3 (8) | 2 (10)
Diarrhea (Gastrointestinal disorders) | 6 (12) | 11 (27)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (10) | 3 (7)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (4) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (4) | 7 (22)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (15)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (12)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 17 (101) | 17 (77)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (12) | 8 (18)
Alkaline phosphatase increased (Investigations) | 2 (22) | 5 (14)
Aspartate aminotransferase increased (Investigations) | 5 (12) | 6 (12)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Cholesterol high (Investigations) | 2 (16) | 1 (3)
Creatinine increased (Investigations) | 2 (17) | 3 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 5 (10) | 3 (5)
GGT increased (Investigations) | 0 (0) | 2 (4)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (44) | 10 (32)
Neutrophil count decreased (Investigations) | 12 (68) | 12 (43)
Platelet count decreased (Investigations) | 8 (26) | 3 (8)
White blood cell decreased (Investigations) | 15 (82) | 17 (65)
Anorexia (Metabolism and nutrition disorders) | 4 (8) | 4 (9)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (33) | 2 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (15) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 1 (7) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (6)
Restlessness (Psychiatric disorders) | 1 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (5)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (10) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (53) | 4 (21)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (14) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 6 (25)
Hypertension (Vascular disorders) | 1 (13) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT02657928/Prot_SAP_000.pdf